CLINICAL TRIAL: NCT02851849
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of Safety and Efficacy of LGD-6972 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LGD-6972 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L6972-04
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LGD-6972-5 mg (Active Comparator): 5 mg LGD-6972 QD
  Interventions: Drug: LGD-6972-5 mg
- LGD-6972-10 mg (Active Comparator): 10 mg LGD-6972 QD
  Interventions: Drug: LGD-6972-10 mg
- LGD-6972-15 mg (Active Comparator): 15 mg LGD-6972 QD
  Interventions: Drug: LGD-6972-15 mg
- Placebo (Placebo Comparator): Placebo QD
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LGD-6972-5 mg — 5 mg LGD-6972 QD
  Other Names: LGD-6972 sodium salt capsules
  Arms: LGD-6972-5 mg
Drug: LGD-6972-10 mg — 10 mg LGD-6972 QD
  Other Names: LGD-6972 sodium salt capsules
  Arms: LGD-6972-10 mg
Drug: LGD-6972-15 mg — 15 mg LGD-6972 QD
  Other Names: LGD-6972 sodium salt capsules
  Arms: LGD-6972-15 mg
Other: Placebo — Placebo QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the change from baseline in hemoglobin A1c (HbA1c) during 12 weeks of treatment with 3 dose levels of LGD-6972 compared to placebo in subjects with Type 2 Diabetes Mellitus (T2DM)

DETAILED DESCRIPTION:
This will be a 12-week, randomized, double-blind, placebo-controlled, 4-arm, parallel group, multi-center study to evaluate the safety and efficacy of LGD-6972 in subjects with T2DM inadequately controlled on metformin monotherapy (a stable [≥12 weeks], daily dose of ≥1000mg at randomization). Subjects with T2DM will be treated with one of 3 dose levels of LGD-6972 (5 mg, 10 mg, or 15 mg) or placebo once daily (QD) for 12 weeks. Randomization will be stratified by HbAlc ≤8.5% or >8.5% at the Placebo Lead-in Visit.

Qualified subjects who require adjustment or stabilization of their metformin dose will participate in a run-in period of up to 12 additional weeks prior to randomization. Subjects will have the option to participate in an oral glucose tolerance test (OGTT) at baseline and end of treatment for assessment of exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects must be surgically sterile (hysterectomy or bilateral oophorectomy or bilateral tubal ligation), or naturally post-menopausal for at least 12 months and with a follicle stimulating hormone (FSH) level in the post-menopausal range (if not taking hormone replacement therapy)
2. Male subjects must either have a vasectomy or agree that they and any female partners will use 2 acceptable forms of contraception, one of which must be a condom, until 30 days after the last dose of study drug. Other acceptable forms of contraception include hormonal contraceptives that have been at stable dose for 12 weeks prior to randomization, intrauterine device, Depo-Provera®, Norplant® System Implants, bilateral tubal ligation, bilateral oophorectomy, hysterectomy, and contraceptive sponge, foam, or jelly. Also, male subjects must not donate sperm during the study and for 30 days after the last dose of study drug
3. Willing and able to provide written informed consent
4. Diagnosis of T2DM according to American Diabetes Association criteria
5. Currently on stable metformin or metformin extended-release therapy (unchanged dose [minimum daily dose of 1000 mg] for ≥12 weeks prior to screening)
6. Subjects must have an HbA1c value of ≥7.0% to ≤10.5%
7. Subjects must have a fasting plasma glucose of ≤260 mg/dL
8. Subjects must have a body mass index (BMI) between 25 kg/m2 and 40 kg/m2, inclusive, and must weigh more than 45 kg

Exclusion Criteria:

1. History of type 1 diabetes mellitus or history of diabetic ketoacidosis or persistent hypoglycemia or hypoglycemia unawareness
2. Women of childbearing potential, lactating, or has a positive pregnancy test
3. History or presence of alcoholism or drug abuse within 2 years prior to screening
4. Unwilling to comply with study restrictions, including restrictions on strenuous exercise
5. Presence of any of the following conditions: renal impairment (defined as history or estimated glomerular filtration rate at screening of <45 mL/min using the Modification of Diet in Renal Disease equation), diabetic proliferative retinopathy, severely symptomatic diabetic neuropathy requiring treatment, diabetic gastroparesis, active liver disease (other than asymptomatic nonalcoholic fatty liver disease), cirrhosis, symptomatic gall bladder disease, or pancreatitis
6. Serum triglyceride level > 400 mg/dL at screening
7. Liver transaminase levels (AST or ALT) >150% ULN, total bilirubin >2 ULN, or creatine kinase (CK) levels > 3 × ULN at screening
8. History or evidence of clinically significant cardiovascular, pulmonary, renal, endocrine (other than T2DM), hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease or surgical intervention (eg, bariatric surgery) or allergic conditions (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
9. Myocardial infarction, unstable angina, arterial revascularization, stroke, symptomatic peripheral artery disease, deep vein thrombosis, New York Heart Association Functional Class III or IV heart failure, or transient ischemic attack within 6 months prior to screening
10. History of malignant hypertension or a recent history of uncontrolled high blood pressure or at screening has a seated systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after at least a 5 minute rest. Blood pressure is determined as the mean of triplicate measurements collected at 2- minute intervals after the subject has been sitting quietly for at least 5 minutes. Therapy for hypertension (beta blockers excluded) that has been stable for at least 8 weeks prior to screening is permitted
11. Arm size in excess of the maximum limit of the largest cuff provided with the study blood pressure monitor
12. History of malignancy (except adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ) within 5 years prior to screening
13. History or evidence of QT prolongation or clinically significant QT prolongation (QTcF >450 msec) at screening, or other significant ECG findings at screening that may place the subject at increased risk by participating in the study
14. Treatment with any type of insulin (injected or inhaled) for > 6 consecutive days within 6 months prior to screening or any insulin therapy within 12 weeks prior to screening
15. Treated with peroxisome proliferator-activated receptor-gamma agonists (thiazolidinediones [TZDs]), incretin therapy (GLP-1 agonists). or amylin mimetics within 12 weeks prior to screening
16. Taking any of the following prohibited medications

    * Antidepressants, antipsychotics, anti-epileptics, hormone replacement therapies (estrogen, progestin), testosterone therapies, and thyroid replacement medications that are not at a stable dose for at least 12 weeks prior to screening
    * Lipid-modifying medications and anti-hypertensive medications that have not been at a stable dose for at least 8 weeks prior to the Screening Visit (excluding bile acid sequestrants, ezetimibe, and beta blockers, which are prohibited
    * Over-the-counter herbal medications and supplement (aside from once daily multivitamins)
17. Treatment with systemic corticosteroids, which must be discontinued at least 4 weeks prior to screening. Note: Inhaled, intraarticular, intranasal and topical corticosteroids are permitted
18. Currently treated with weight-loss medications. These must be discontinued ≥12 weeks prior to screening
19. History or evidence of intravenous illicit drug use, active hepatitis B virus (HBV), hepatitis C virus (HCV), and/or human immunodeficiency virus (HIV) infection
20. Known hypersensitivity or idiosyncratic reaction to glucagon receptor (GCGR) antagonists or LGD-6972
21. Participation in another interventional clinical trial within 30 days prior to dosing or treatment with an investigational product with 14 days or 5 half-lives of the Screening Visit (whichever is longer)
22. Donated ≥ 450 mL of blood within 56 days of screening or has donated blood products within 30 days of screening
23. Inability to comply with study procedures or to adhere to study-required restrictions

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline in HbA1C | Baseline to Weeks 2,4,8
Change from baseline in fasting glucose | Baseline to Weeks 2,4,8 and 12
Change from baseline values for fasting glucagon | Baseline to Weeks 2,4,8 and 12
Change from baseline values for fasting GLP-1 (total and active) | Baseline to Weeks 2,4,8 and 12
Change from baseline values for fasting insulin | Baseline to Weeks 2,4,8 and 12
Change from baseline values for fasting lipids (total, LDL, and HDL cholesterol and triglycerides) | Baseline to Weeks 2,4,8, and 12
Change from baseline in blood pressure (systolic and diastolic) | Baseline to Weeks 2,4,8, and 12
Change from baseline in body weight | Baseline to Weeks 2,4,8 and 12

OTHER OUTCOMES:
Exploratory Objective - Change from baseline from an Oral Glucose Tolerance Test (area under the curve for glucose, glucagon, insulin, C-peptide, and total and active GLP-1) | Baseline, 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keith Marschke, Ph.D., Study Director — Ligand Pharmaceuticals
Locations (27):
- United States (27):
  - Tuscumbia, Alabama
  - Chandler, Arizona
  - Surprise, Arizona
  - Huntington Park, California
  - Los Angeles, California
  - Montclair, California
  - North Hollywood, California
  - San Diego, California
  - Denver, Colorado
  - Brooksville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Hopewell Junction, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Franklin, Ohio
  - Munroe Falls, Ohio
  - Summerville, South Carolina
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - Katy, Texas
  - Manassas, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pettus JH, D'Alessio D, Frias JP, Vajda EG, Pipkin JD, Rosenstock J, Williamson G, Zangmeister MA, Zhi L, Marschke KB. Efficacy and Safety of the Glucagon Receptor Antagonist RVT-1502 in Type 2 Diabetes Uncontrolled on Metformin Monotherapy: A 12-Week Dose-Ranging Study. Diabetes Care. 2020 Jan;43(1):161-168. doi: 10.2337/dc19-1328. Epub 2019 Nov 6. PMID 31694861